CLINICAL TRIAL: NCT00118131
Title: Phase II Study of Weekly Docetaxel Together With Weekly Cisplatin in Chemotherapy-Naive Patients With Stage IV or Select Stage IIIB (Malignant Effusion) Non-Small Cell Lung Cancer
Brief Title: Docetaxel and Cisplatin in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000433488; P30CA072720 (NIH); CINJ-030302 (Other: Cancer Institute of New Jersey); CINJ-NJ1503 (Other: Cancer Institute of New Jersey)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel and Cisplatin (Experimental): A cycle is defined as an interval of 28 days.
  Docetaxel, 35 mg/m2 per day on Days 1, 8 and 15 (total dose for this cycle = 105 mg/m2).
  Cisplatin, 25 mg/m2 per day on Days 1, 8 and 15 (total dose for this cycle = 75 mg/m2).
  Docetaxel is always to be given prior to cisplatin on Days 1, 8 and 15.
  Interventions: Drug: cisplatin; Drug: docetaxel

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with cisplatin works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of docetaxel and cisplatin, as measured by tumor response rate, in patients with chemotherapy-naïve stage IIIB or IV non-small cell lung cancer.

Secondary

* Determine the duration of response in patients treated with this regimen.
* Determine time to disease progression in patients treated with this regimen.
* Determine the 1-year survival rate in patients treated with this regimen.
* Determine the median survival time in patients treated with this regimen.
* Correlate aneuploidy (as determined by DNA histograms) and immunohistochemical expression of stathmin, Aurora-A, and survivin with response in patients treated with this regimen.

OUTLINE: This is an open-label, nonrandomized, multicenter study.

Patients receive docetaxel IV over 1 hour and cisplatin IV over 1 hour once on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 76 patients will be accrued for this study within 13-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer, meeting 1 of the following stage criteria:

  * Stage IIIB disease with malignant pericardial or malignant pleural effusions, as indicated by 1 of the following:

    * Positive cytology
    * Exudative effusion AND lactic dehydrogenase (LDH) > 200 IU with effusion/serum LDH ratio ≥ 0.6
  * Stage IV disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques OR > 10 mm by spiral CT scan
* Brain metastases allowed provided they have been irradiated AND are radiographically stable for ≥ 28 days after the completion of radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* AST and ALT normal
* Bilirubin normal

Renal

* Creatinine clearance ≥ 50 mL/min

Immunologic

* No known HIV positivity
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No clinically significant active infection

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception before, during, and for 4 weeks after completion of study treatment
* No other primary malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious systemic disorder that would preclude study participation
* No other condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior antibody-based therapy that targets growth factor pathways (e.g., epidermal growth factor receptor [EGFR]) allowed provided there is disease progression during therapy and patient has recovered
* No concurrent immunotherapy
* No concurrent prophylactic colony-stimulating factors
* No concurrent interleukin-11

Chemotherapy

* No prior cytotoxic chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy for the malignancy

Radiotherapy

* See Disease Characteristics
* More than 28 days since prior radiotherapy and recovered
* No prior radiotherapy to ≥ 25% of the bone marrow
* No prior radiotherapy to sites of measurable disease unless there is documented tumor progression after completion of radiotherapy
* No concurrent radiotherapy

Surgery

* No concurrent surgery for the malignancy

Other

* More than 3 weeks since prior investigational drugs
* Prior oral small molecule drug therapy that targets growth factor pathways (e.g., EGFR) allowed provided there is disease progression during therapy and patient has recovered
* No other concurrent investigational or commercial agents or therapies for the malignancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Aisner, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (13):
- United States (13):
  - Central Jersey Oncology Center, PA - East Brunswick, East Brunswick, New Jersey
  - JFK Medical Center in Edison, Edison, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - UMDNJ - University Hospital, Newark, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center) and 4 affiliate community hospitals part of the Cancer Institute of New Jersey Oncology Group from December 2003 through February 2008.
Period: Overall Study
Arm/Group | Docetaxel and Cisplatin
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and Cisplatin
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response Rate
Description: Patients experiencing complete or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: 7 years
Population: Analysis was performed on the first 47 patients. Study was Terminated before 2 of the patients met the pre-specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel and Cisplatin
Number analyzed (Participants) | 47
percentage of participants | 21

2. Secondary Outcome: Time to Progressive Disease
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 8 years
Population: Analysis was performed on the first 47 patients . Study was Terminated before 2 of the patients met the pre-specified time point.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and Cisplatin
Number analyzed (Participants) | 47
months | 3.38 [2.3 to 5.8]

3. Secondary Outcome: 1-year Survival Rate
Time Frame: 1 year
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel and Cisplatin
Number analyzed (Participants) | 47
percentage of participants | 38

4. Secondary Outcome: Median Survival Time
Time Frame: 10 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and Cisplatin
Number analyzed (Participants) | 47
months | 9.1 [5.8 to 14.9]

ADVERSE EVENTS:
Time Frame: From the start of baseline to the end of the study up to 5 years.
Arm/Group | Docetaxel and Cisplatin
All-Cause Mortality (participants affected / at risk) | 45/49
Serious Adverse Events (participants affected / at risk) | 18/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Cisplatin (N=49)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 2 (2)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 2 (2)
Hyperglycemia (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Hypomagnesemia (Investigations) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1)
Seizure(s) (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary-Other (Specify, RLL pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary-Other (Specify, respiratory distress) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Thrombosis/embolism - pulmonary embolism (Vascular disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Cisplatin (N=49)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 23 (31)
Nausea (Gastrointestinal disorders) | 19 (26)
Constipation (Gastrointestinal disorders) | 16 (18)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 15 (19)
Anorexia (Gastrointestinal disorders) | 14 (15)
Vomiting (Gastrointestinal disorders) | 9 (12)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 8 (8)
Dyspepsia/heartburn (Gastrointestinal disorders) | 5 (5)
Dehydration (Gastrointestinal disorders) | 5 (5)
Gastrointestinal (Gastrointestinal disorders) | 5 (5)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (27)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Nail changes (Skin and subcutaneous tissue disorders) | 3 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 25 (29)
Weight loss (General disorders) | 5 (6)
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 3 (4)
Neuropathy-sensory (Nervous system disorders) | 12 (16)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 7 (8)
Insomnia (Nervous system disorders) | 6 (9)
Dizziness/lightheadedness (Nervous system disorders) | 5 (5)
Mood alteration-depression (Psychiatric disorders) | 5 (5)
Neuropathy - motor (Nervous system disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 19 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (16)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pain (General disorders) | 10 (13)
Bone pain (General disorders) | 4 (4)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 3 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 10 (12)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 5 (7)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (7)
Hemoglobin (Blood and lymphatic system disorders) | 4 (6)
Thrombosis/embolism (Vascular disorders) | 4 (4)
Edema (Vascular disorders) | 9 (11)
Creatinine (Renal and urinary disorders) | 4 (7)
Renal/Genitourinary (Renal and urinary disorders) | 4 (5)
Hypomagnesemia (Investigations) | 6 (6)
Hyponatremia (Investigations) | 5 (5)
Hypokalemia (Investigations) | 4 (4)
Hyperglycemia (Investigations) | 3 (6)
Ocular/Visual (Eye disorders) | 4 (4)
Tearing (watery eyes) (Eye disorders) | 4 (5)
Infection without neutropenia (Infections and infestations) | 5 (6)
Hemoptysis (Blood and lymphatic system disorders) | 4 (4)
Palpitations (Cardiac disorders) | 3 (3)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 3 (3)
Hypoalbuminemia (Hepatobiliary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes